CLINICAL TRIAL: NCT03790241
Title: In Vivo Biomechanical Analysis of the Practitioner's Motion During a Peripheral Venous Catheter Insertion
Acronym: ABGPVVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0533; 2018-A02895-50 (Other: ANSM Number)
Record Dates: First submitted 2018-12-06; First posted 2018-12-31 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: catheter insertion; puncture; skin; vein; palpation; motion tracking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Young males of normal corpulence (Experimental): Insertion of a catheter to people ageg between 18 and 25; IBM between 18,5 and 25
  Interventions: Procedure: insertion of a catheter
- Young females of normal corpulence (Experimental): Insertion of a catheter to people ageg between 18 and 25; IBM between 18,5 and 25
  Interventions: Procedure: insertion of a catheter
- Aged males of normal corpulence (Experimental): Insertion of a catheter to people ageg between 60 and 75; IBM between 18,5 and 25
  Interventions: Procedure: insertion of a catheter
- Aged females of normal corpulence (Experimental): Insertion of a catheter to people ageg between 60 and 75; IBM between 18,5 and 25
  Interventions: Procedure: insertion of a catheter
- Obese young males (Experimental): Insertion of a catheter to people ageg between 18 and 25; superior or equal to 30
  Interventions: Procedure: insertion of a catheter
- Obese young females (Experimental): Insertion of a catheter to people ageg between 18 and 25; superior or equal to 30
  Interventions: Procedure: insertion of a catheter
- Obese aged males (Experimental): Insertion of a catheter to people ageg between 60 and 75; IBM superior or equal to 30
  Interventions: Procedure: insertion of a catheter
- Obese aged females (Experimental): Insertion of a catheter to people ageg between 60 and 75; IBM superior or equal to 30
  Interventions: Procedure: insertion of a catheter

INTERVENTIONS:
Procedure: insertion of a catheter — Analysis the palpation and perforation motion performed by the practitioner during the insertion of a catheter while measuring the loads applied on the skin and the veins

SUMMARY:
The aim of this study is to analyze the palpation and perforation motion performed by the practitioner during the insertion of a catheter while measuring the loads applied on the skin and the veins.

These experimental measures will be used for the design of a more realistic peripheral venous catheter insertion simulator in order to better prepare healthcare students for their first in vivo venous puncture.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteer
* Aged between 18-25 yo or 60-75 yo
* IBM between 18,5-25 or superior or equal to 30
* Cognitive level compatible with oral communication, respect of safety instructions and understanding of realized acts
* Signed the study agreement

Exclusion Criteria:

* Individuals displaying coagulation disorders
* Individuals displaying skin lesions, scars or areteriovenous fistula on the ventral side of the forearm
* Individuals displaying a high infection risk
* Women that have been subject to a lymph node dissection on a malignant breast tumor
* Individuals not able to express their consent
* Individuals having a hierarchical link with the persons conducting this study
* Individuals currently participating to another research which includes an exclusion period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Punctures forces of the skin and veins measured by an instrumented syringue | Day 0 (at intervention)
  According to the literature, puncture forces of soft tissues are decomposed as a summation of stiffness forces, friction forces and cutting forces. In the case of this study, an instrumented syringe has been designed to measure the puncture force in function of time. This device includes a miniature1-axis load sensor. The catheters can be easily removed thanks to a conical fitting which is directly connected to the load sensor to obtain the forces when inserting and withdrawing the catheter.
  The primary sought measures are the peak force occurring when penetrating the skin and the vein as well as the friction forces when withdrawing the catheter from the vein.
Needle velocity during perforation measured by a flexible piezoresistive sensor | Day 0
  In order to obtain the load applied by the practitioner to locate the vein to puncture, a flexible piezoresistive sensor is placed to the practitioner's fingertip with double side tape The sensor is linked to its acquisition module which is connected via Wi-Fi to a computer.
  In order to not disturb the motion of the practitioner, the module if fixed with a sport armband to the forearm.
  The primary sought measure is the curve force in function of time.
Needle insertion angle during perforation measured by digital image correlation | Day 0
  obtained thanks to digital image correlation which consists of tracking sights with two high speed cameras. Thus, sights will be placed on the side of the palpating finger and instrumented syringe.
Loads applied by the palpating finger to locate the vein to puncture, measured by digital image correlation | Day 0
  obtained thanks to digital image correlation which consists of tracking sights with two high speed cameras. Thus, sights will be placed on the side of the palpating finger and instrumented syringe.
Spatial displacement of the palpating finger measured by digital image correlation | Day 0
  obtained thanks to digital image correlation which consists of tracking sights with two high speed cameras. Thus, sights will be placed on the side of the palpating finger and instrumented syringe.

SECONDARY OUTCOMES:
Age | Day 0
  to evaluate the Influence of age regarding the puncture forces
Sex | Day 0
  to evaluate the Influence of sex regarding the puncture forces
Weight | Day 0
  to measure body mass index BMI and evaluate the its Influence of regarding the puncture forces
Height | Day 0
  to measure body mass index BMI and evaluate the its Influence of regarding the puncture forces

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Biomechanics and Impact Mechanics - Centre Hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torossian K, Ottenio M, Brulez AC, Lafon Y, Viste A, Attali P, Benayoun S. Biomechanical analysis of practitioner's gesture for peripheral venous catheter insertion. Med Eng Phys. 2021 Apr;90:92-99. doi: 10.1016/j.medengphy.2021.03.001. Epub 2021 Mar 4. PMID 33781485